CLINICAL TRIAL: NCT05640362
Title: Efficacy of Natural Enzymes Mouthwash: a Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: UKM PPI/111/8/JEP-2016-582
Record Dates: First submitted 2022-11-28; First posted 2022-12-07 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-11

CONDITIONS: Xerostomia; Dry Mouth
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Benzydamine mouthwash (Placebo Comparator)
  Interventions: Other: Benzydamine mouthwash
- Natural enzymes mouthwash (Experimental)
  Interventions: Other: Natural enzymes mouthwash

INTERVENTIONS:
Other: Natural enzymes mouthwash — Natural enzymes mouthwash contains numerous natural protein-enzymes, including lactoferrin, lysozyme, lactoperoxidase, glucose oxidase. These active ingredients were proposed to render this mouthwash to act as salivary substitutes by reinforcing the functions of available saliva, hence reinforcing the immune system in the oral cavity. It was expected to relieve the symptoms in xerostomia patients, and even more if the patients have salivary flow reduction by improving the functions of the limited amount of saliva. The potential mechanisms of action of the mouthwash to treat xerostomia may be related to: (1) lubrication effects to wet the oral mucosal surfaces; (2) antimicrobial properties that will reduce risks of mucosal irritation by infections; (3) absence of alcohol in the mouthwash Subjects were instructed to rinse with the mouthwash 4 times per day at a specific period, for 2 weeks.
  Other Names: Oral7 mouthwash
  Arms: Natural enzymes mouthwash
Other: Benzydamine mouthwash — Subjects were instructed to rinse with the mouthwash 4 times per day at a specific period, for 2 weeks.
  Other Names: Difflam mouthwash
  Arms: Benzydamine mouthwash

SUMMARY:
The goal of this clinical is to assess the efficacy of natural enzymes mouthwash in the treatment of xerostomia (dry mouth). The main questions it aims to answer are: (1) the efficacy of natural enzymes mouthwash in the symptomatic treatment of xerostomia; and (2) the response of xerostomia patients towards natural enzymes mouthwash. Participants were given a mouthwash to be used. Intervention group received natural enzymes moisturising mouthwash, while control group received benzydamine mouthwash. Mouthwashes were repacked, labelled with specific code and were given to participants by third-party. Subjects were instructed to rinse with the mouthwash 4 times per day at a specific period, for 2 weeks. Data were compared within each arm before and after using the mouthwashes; and between both arms after using the mouthwashes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above,
* complained of dry mouth (xerostomia), and
* taking nutrition orally

Exclusion Criteria:

* patients who had been using mouthwash for xerostomia in the past 1 week,
* unable to provide saliva samples,
* unable to chew paraffin wax for stimulated saliva,
* patients with oral motor function deficits, and
* those with severe cognitive deterioration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2017-03-09 (Actual); Study Completion 2017-03-24 (Actual)

PRIMARY OUTCOMES:
Changes in symptoms | At Day 0 and Day 14 of intervention
  Symptoms of xerostomia assessment using Xerostomia Inventory

SECONDARY OUTCOMES:
Changes in clinical signs | At Day 0 and Day 14 of intervention
  Signs of xerostomia assessment using Clinical Oral Dryness Score (CODS)
Salivary flow rate | At Day 0 and Day 14 of intervention
  Resting and stimulated salivary flow rate

CONTACTS AND LOCATIONS:
Overall Officials: Rifqah Nordin, MClinDent, Principal Investigator — National University of Malaysia
Locations (1):
- Faculty of Dentistry, Universiti Kebangsaan Malaysia, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiam TL, Choo J, Ashar A, Hussaini HM, Rajandram RK, Nordin R. Efficacy of natural enzymes mouthwash: a randomised controlled trial. Clin Oral Investig. 2024 Apr 19;28(5):259. doi: 10.1007/s00784-024-05658-7. PMID 38639763